CLINICAL TRIAL: NCT04664673
Title: Effect of the Intensive Intervention "Hand-Arm Bimanual Intensive Therapy Including Lower Extremities" (HABIT-ILE) in Chronic (> 6 Months) Adults With Acquired Brain Damage (Stroke)
Brief Title: HABIT-ILE in Adults With Chronic Stroke (HABIT-ILE Stroke)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: University Hospital of Mont-Godinne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B403201316810h
Record Dates: First submitted 2020-12-02; First posted 2020-12-11 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Allocation
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE (Experimental): HABIT-ILE (Hand-Arm Bimanual Intensive Therapy Including Lower Extremities) intervention during two weeks adapted for adults stroke survivors
  Interventions: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)
- Regular care (Active Comparator): Usual customary treatment for adults stroke survivors during two weeks
  Interventions: Behavioral: Regular care

INTERVENTIONS:
Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) — motor learning-based, intensive therapy originally developed for hemiplegic children.
  Other Names: HABIT-ILE Stroke
  Arms: HABIT-ILE
Behavioral: Regular care — customary or usual treatment given to any adult stroke survivor
  Other Names: Usual care
  Arms: Regular care

SUMMARY:
Using a randomized controlled trial design, the possible changes induced by the intensive treatment program "Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)" will be studied in functional, everyday life activities and neuroplastic assessment of adults with chronic stroke.

DETAILED DESCRIPTION:
Using a randomized controlled trial design, the possible changes in neuroimaging, motor function, motor learning and everyday life activities of adults with chronic stroke (> 6 months) after participating of the intensive treatment programme "Hand-arm Bimanual Intensive Therapy Including Lower Extremities" (HABIT-ILE) will be studied. Changes, scored by participants in case of questionnaires and by experts in the case of tests, will be observed comparing participants after their regular care/treatment and after receiving HABIT-ILE. Motor function, learning and daily life activities will be correlated with neuroplastic changes.

ELIGIBILITY:
Inclusion Criteria:

* hemiparetic patient with a chronic stroke (over 6 months of evolution)
* age 40 to 90 years old inclusive
* ability to follow instructions and complete testing according to the age.

Exclusion Criteria:

* alcohol/drug abuse
* pregnancy
* major cognitive impairment interfering with the study (severe aphasia, psychiatric conditions)
* uncontrolled health issues (cardiac/renal failure)
* contraindications to perform MRI assessments (Metal implants, etc.)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes on the Adult Assisting Hand Assessment Stroke (Ad-AHA Stroke) | baseline, 3 weeks and 13 weeks after baseline
  This assessment is an observation-based instrument assessing the effectiveness of the spontaneous use of the affected hand when performing bimanual activities in adults post stroke scored in a logit based 0-100 AHA-unit scale (higher score indicate higher ability)

SECONDARY OUTCOMES:
Changes on speed/accuracy trade-off during a bimanual reaching task (bi-SAT) | baseline, 3 weeks and 13 weeks after baseline
  By using the Rehabilitation Robot System (REAplan®), we calculate the bi-SAT through mathematical computation
Changes on force during a bimanual reaching task (bi-Force) | baseline, 3 weeks and 13 weeks after baseline
  By using the REAplan® robot, we calculate the bimanual forces and forces exerted in the wrong direction by each arm (Newtons)
Changes on bimanual coordination during a bimanual reaching task (bi-CO) | baseline, 3 weeks and 13 weeks after baseline
  By using the REAplan® robot, we calculate the phase coherence between speeds of both arms
Changes on bimanual smoothness during a bimanual reaching task (bi-smoothness) | baseline, 3 weeks and 13 weeks after baseline
  By using the REAplan® robot, we calculate the Spectral Arc Length (SPARC) of the movement (unitless)
Changes on errors during a bimanual reaching task (bi-error) | baseline, 3 weeks and 13 weeks after baseline
  By using the REAplan® robot, we calculate the amount of errors while performing the bimanual task (measured in centimeters or degrees)
Changes in finger force tracking dexterity | baseline, 3 weeks and 13 weeks after baseline
  By using a finger force manipulandum (DEXTRAIN), which records the forces (in Newtons) applied by the fingers on pistons, we calculate the ability to control and release the force applied by the fingers during a tracking task.
Changes in multifinger tapping dexterity | baseline, 3 weeks and 13 weeks after baseline
  By using the DEXTRAIN, we assess the independent finger movements while simultaneous tapping with different finger configurations (two fingers or one finger) in response to visual instructions during a finger tapping task. The percentage of errors are considered.
Changes in cortical thickness of the brain's gray matter | baseline, 3 weeks and 13 weeks after baseline
  Regional brain cortical thickness is acquired from high resolution 3D T1-weighted structural imaging data. For each investigated region, mean cortical metrics (in millimeters) are assessed between the pial surface and the white/grey boundary.
Changes in Fractional Anisotropy (FA) of the corticospinal tract from the motor cortex to the cerebellar peduncle | baseline, 3 weeks and 13 weeks after baseline
  FA is a scalar value (no unit) between 0 and 1 that describes the degree of anisotropy of white matter water molecules. It is measured non-invasively via brain MRI using diffusion tensor imaging (DTI), a modality of Diffusion-Weighted Imaging (DWI). Increased values indicate a higher directionality of the tissue structure.
Changes on the Axial, Radial and Mean Diffusivity (AD, RD, MD) of the corticospinal tract from the motor cortex to the cerebellar peduncle | baseline, 3 weeks and 13 weeks after baseline
  AD, RD and MD are values ranging from 0 to 3.10-3 [mm2/s] that describe the degree of axial, radial and mean molecular diffusion of white matter water molecules. It is measured non-invasively via brain MRI using diffusion tensor imaging (DTI), a modality of Diffusion-Weighted Imaging (DWI). An increased MD can be considered to be an indicator of white matter damage.
Changes on the metrics of the corticospinal tract from the motor cortex to the cerebellar peduncle using the NODDI model | baseline, 3 weeks and 13 weeks after baseline
  The orientation dispersion index (ODI), intracellular volume fraction (ICVF) and the fraction of the isotropic compartment (ISOF) are scalar values ranging from 0 to 1 (no units) that describe the orientation of neural fibers, and the volume fraction of the intracellular and isotropic compartment. It is measured non-invasively via brain MRI using the Neurite Orientation Dispersion and Density Imaging (NODDI) model combined with a Diffusion-Weighted Imaging (DWI) sequence. The results reflects the overall coherence of the fibers, with zero representing highly coherent structures, hence less dispersion of the fibers.
Changes on the metrics of the corticospinal tract from the motor cortex to the cerebellar peduncle using the DIAMOND model | baseline, 3 weeks and 13 weeks after baseline
  By representing each voxel of the brain as the sum of multiple compartments (representing either a neural fiber population or an isotropic diffusion), the volume fraction and the heterogeneity of each compartment can be estimated. These metrics (ranging from 0 to 1, no unit) are measured non-invasively via brain MRI using the Distribution of 3D Anisotropic Microstructural environments in Diffusion-compartment imaging (DIAMOND) model combined with a Diffusion-Weighted Imaging (DWI) sequence. The results reflects the overall heterogeneity of the fibers, with zero representing more homogeny structures, hence less dispersion of the fibers.
Changes in resting-state functional connectivity | baseline, 3 weeks and 13 weeks after baseline
  Resting-state functional magnetic resonance imaging (rs-fMRI) evaluates the regional interactions that occur during the resting or task-negative state. The magnitude of the brain activation during rs-fMRI will be assessed
Changes in brain white matter microstructure (WM-μs) using the Microstructure Fingerprinting model | baseline, 3 weeks and 13 weeks after baseline
  Using a multiple-compartment approach, the signal obtained from a voxel can be estimated as the sum of multiple fiber populations, each presenting a specific fraction ('frac', ranging from 0 to 1, no unit), fiber volume fraction ('fvf', ranging from 0 to 1, no unit) and diffusivity ('diff', in [mm2/s]). On top of those fiber populations, isotropic compartments can also be represented with a specific fraction (frac) and diffusivity (diff). These metrics are measured non-invasively via brain MRI using the Microstructure Fingerprinting model combined with a Diffusion-Weighted Imaging (DWI) sequence.
Changes in upper extremities sensorimotor functions assess by the Fugl-Meyer Assessment (FMA-UE) | baseline, 3 weeks and 13 weeks after baseline
  The FMA-UE assess reflex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia. Maximum score is 66 points (Higher scores indicates better functioning levels)
Changes in upper extremities motor functions assess by the Wolf Motor Function Test (WMFT) | baseline, 3 weeks and 13 weeks after baseline
  The WMFT measures quantitative motor ability through 17 timed and functional tasks. Uses a 6-point ordinal scale (from 0= "does not attempt with the involved arm" to 5= "arm does participate; movement appears to be normal"). Maximum score is 75 (Higher scores indicates better functioning levels)
Changes in unimanual dexterity assessed by the Box & Block test (BBT) | baseline, 3 weeks and 13 weeks after baseline
  The BBT assess unimanual dexterity by quantifying the maximum of wooden blocks transferred from one space to the other during 1 minute (Higher scores indicate better performance)
Changes in the Six Minutes' Walk Test (6MWT) | baseline, 3 weeks and 13 weeks after baseline
  The 6MWT assess endurance while walking 6 minutes without pause. More distance walked (in meters) indicate better performance
Changes in Canadian Occupational Performance Measure (COPM) | baseline, 3 weeks and 13 weeks after baseline
  In this interview, patients set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the patient's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10)
Changes in the Stroke Impact Scale (SIS) | baseline, 3 weeks and 13 weeks after baseline
  Self-reported questionnaire assessing multidimensional repercussions of the Stroke (strength, hand function, daily life activities, mobility, communication, emotion, memory, thinking and participation). Domains are scored on a metric of 0 to 100 (higher scores indicate better self-reported health)
Changes in activities of daily living assessed by ACTIVLIM-Stroke Questionnaire | baseline, 3 weeks and 13 weeks after baseline
  The ACTIVLIM-Stroke questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or lower extremities through 20 items specific to patients after stroke. It ranges from - 6 to +6 logits (higher score means better performance).
Changes in activities of daily living assessed by ABILHAND Questionnaire | baseline, 3 weeks and 13 weeks after baseline
  The ABILHAND questionnaire specific to patients with chronic stroke measures a patient's manual ability to manage daily activities that require the use of the upper extremities, whatever the strategies involved, through 23 items. It ranges from -6 to +6 logits (higher score means better performance).
Changes in the modified Rankin Scale (mRS) for neurologic disability | baseline, 3 weeks and 13 weeks after baseline
  mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The 6 levels of disability goes from 0 ("no disability/no symptoms") to 5 ("disability requiring constant care for all needs"), being 6 "death".
Changes in visual neglect assessed by the Bells Test | baseline, 3 weeks and 13 weeks after baseline
  The Bells Test is a cancellation test that allows for a quantitative and qualitative assessment of visual neglect in the near extra personal space. The patient score is based on the amount of time they take to complete the task, and the number of correct items (35 bells) they identify.
Changes on the visuospatial short term working memory assessed by the "Corsi block-tapping test" | baseline, 3 weeks and 13 weeks after baseline
  The test requires the patient to observe and then repeat in order a sequence of blocks "tapped". The task starts with a sequence of 2 blocks and gradually increases in length up to nine blocks. The test measures both the number of correct sequences and the longest sequence remembered. This number is known as the "Corsi Span", and averages about 5 for normal human subjects.
Changes in the Montreal Cognitive Assessment (MoCA) test | baseline, 3 weeks and 13 weeks after baseline
  The MoCA is a brief screening instrument originally designed to identify mild cognitive impairments in elderly patients attending a memory clinic. MoCA evaluates different domains (visuospatial abilities, executive functions, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space) having a total of 30 points (higher scores indicate better self-reported health)
Changes in inhibitory control assessed by the Stroop Color and Word Test (SCWT) | baseline, 3 weeks and 13 weeks after baseline
  The SCWT is extensively used to assess the ability to inhibit cognitive interference occurring when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. The reaction time and the amount of errors are measured during incongruent and congruent tasks (lower reaction times and less errors indicates better performance).
Changes in executive functions assessed by the Trail Making Test (TMT) | baseline, 3 weeks and 13 weeks after baseline
  The TMT provides information on visual search, scanning, speed of processing, mental flexibility and executive functions using two subtasks, link numbers in increasing order and link letters and numbers in increasing order. The reaction time and the amount of errors are measured during the subtasks (lower reaction times and less errors indicates better performance).
Changes in the Wechsler Adult Intelligence Scale (WAIS-III) | baseline, 3 weeks and 13 weeks after baseline
  The WAIS-III provided scores for Verbal intelligence quotient (IQ), Performance IQ, and Full Scale IQ, along with four secondary indices (Verbal Comprehension, Working Memory, Perceptual Organization, and Processing Speed). The six Verbal Scale (Vocabulary, Similarities, Arithmetic, Digit Span, Information, and Comprehension) and five Performance Scale (Picture Completion, Digit Symbol (Coding), Block Design, Matrix Reasoning, and Picture Arrangement) subtests are combined to calculate the Full Scale IQ. After each subtest is scored, raw point totals are converted to scaled scores according to the examinee's age range (mean= 10; standard deviation=3). Sums of scaled scores then are computed separately for the six Verbal Scale subtests, five Performance Scale subtests, and all 11 subtests which constitute the Full Scale. The sums are converted to deviation IQs. The IQs generated have a mean of 100 and a standard deviation of 15 at all age levels.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Vandermeeren, MD,PhD, Principal Investigator — Institute of Neuroscience, UCLouvain; CHU-UCL Namur, Neurology Department, UCLouvain; Yannick Bleyenheuft, PhD, Principal Investigator — MSL-IN Lab, Institute of Neuroscience, UCLouvain
Locations (1):
- Institute of Neuroscience, UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebner-Karestinos D, Gathy E, Carton de Tournai A, Herman E, Araneda R, Dricot L, Macq B, Vandermeeren Y, Bleyenheuft Y. Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) in adults with chronic stroke: protocol of a randomised controlled trial. BMJ Open. 2023 Apr 13;13(4):e070642. doi: 10.1136/bmjopen-2022-070642. PMID 37055214